CLINICAL TRIAL: NCT00537706
Title: Engaging Low-Income Urban Residents in Prioritizing Interventions to Address Socio-Economic Determinants of Health
Brief Title: Choosing Healthful Interventions
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907224; 07-CC-N224
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-10-31

CONDITIONS: Socioeconomic Factors; Low-Income Population; Health Status
Keywords: Socioeconomic Determinants; Health Status; Low-income; Priority-setting; Group Discussion

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will identify what programs, along with traditional healthcare, low-income urban residents would choose to improve their health. The information is intended as a step toward designing public policies aimed at improving the health of low-income populations in the United States.

Residents of Washington, D.C., who are between 18 and 64 years of age and are in a specified income bracket may be eligible for this study.

Participants take part in audio-taped group discussions led by a trained facilitator. During a 3 hour session, participants engage in 4 cycles of choosing benefits. Participants select benefits as follows:

* For themselves individually.
* For their neighborhood.
* For an entire city.
* Once again individually.

DETAILED DESCRIPTION:
BACKGROUND:

There is a growing recognition that health status is only partially a function of health care. Socio-economic determinants of health, particularly income status and education, have significant effects on health status and outcomes. In light of these socio-economic determinants, several governments in the Organization for Economic Cooperation and Development (OECD) are adopting evidence-based policy recommendations for improving the health of their populations. Britain has conducted research that has been path breaking in identifying these determinants of health and in planning to address them. Canada has similar plans.

OBJECTIVE:

The goal of this project is to explore the possibility of designing public policies aimed at improving the health of urban low-income populations in the US. Toward this end, this project will engage health policy experts and low-income residents in an exploratory exercise aimed at designing an affordable, evidence-based intervention program targeted at addressing socio-economic factors and reducing health disparities among low income residents of Washington, DC. A three step process will be carried out:

1. Identification of candidate interventions that have been shown to ameliorate the socio-economic determinants of health, through literature review and consultation with experts;
2. Consideration of a reasonable per capita expenditure for the purpose;
3. Engagement of low-income residents to ascertain their priorities for publicly funding the proposed interventions within the assigned budget.

Several hundred low-income adults recruited from clinical and community settings will participate in this engagement process through small group exercises in which a facilitated discussion will take place using a previously tested group decision tool, REACH (Reaching Economic Alternatives that Contribute to Health). Data pertaining to participants' socio-demographic characteristics, attitudes toward health, and preferences for possible interventions will be collected anonymously. Group discussions will be audio-taped. Data will be analyzed quantitatively and qualitatively to determine preferences for various interventions and their association with socio-demographic characteristics. Participants will be financially compensated with $75 for their participation.

RISKS AND BENEFITS:

Given the anonymous nature of the data collection, we anticipate no risks other than those entailed in discussion of poor health outcomes associated with lack of insurance and low income. Participants may benefit from learning about factors that improve health status.

OUTCOME AND MEANING TO THE FIELD:

Study results will yield information about benefits that are of utmost priority to low income urban residents. This is unique information that may contribute to efforts to find affordable strategies for ameliorating the socio-economic determinants of health for low-income urban population in the US.

ELIGIBILITY:
* INCLUSION CRITERIA:

Low-income male and female adults will be recruited as study participants.

EXCLUSION CRITERIA:

Children 18 years and younger are ineligible.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 442 (Estimated)
Dates: Start 2007-09-21; Study Completion 2011-10-31

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ames, R.N., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- Howard University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Danis M, Lovett F, Sabik L, Adikes K, Cheng G, Aomo T. Low-income employees' choices regarding employment benefits aimed at improving the socioeconomic determinants of health. Am J Public Health. 2007 Sep;97(9):1650-7. doi: 10.2105/AJPH.2006.091033. Epub 2007 Jul 31. PMID 17666702